CLINICAL TRIAL: NCT00156949
Title: An Open-Label, Single-Arm Study to Assess the Safety of Epoetin Alfa Manufactured by a Deep Tank Technology in Subjects With Chronic Kidney Disease Receiving Dialysis
Brief Title: EPO Deep Tank in Dialysis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040268
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Kidney Disease
Keywords: Epogen; Procrit; Chronic Kidney Disease; Anemia Treatment for Dialysis Patients
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Epoetin Alfa

ARMS (1):
- Epoetin alfa DT (Experimental)
  Interventions: Drug: Epoetin alfa DT

INTERVENTIONS:
Drug: Epoetin alfa DT — Receive drug at same frequency and dose as at the time of randomization Change dose by+/- 25% in order to maintain Hb between 11.0 - 13.0 g/dL

SUMMARY:
Subject incidence of adverse events

DETAILED DESCRIPTION:
To determine whether Epoetin alfa manufactured by a roller bottle technology (Epoetin alfa RB) and Epoetin alfa manufactured by a deep tank process (Epoetin alfa DT) have comparable safety profiles when administered to patients with CKD receiving dialysis.

ELIGIBILITY:
Inclusion Criteria: - ≥ 18 years of age - Receiving hemodialysis or peritoneal dialysis - Baseline Hb between 11.0 g/dL and 13.0 g/dL - Currently receiving Epoetin alfa RB ie. EPOGEN or PROCRIT - Transferrin saturation (Tsat) >15.0% Exclusion Criteria: - Currently receiving or ever received treatment with any erythropoietic stimulating protein other than EPOGEN, Procrit and Aranesp. - Uncontrolled hypertension (defined as diastolic blood pressure >110 mmHg or systolic BP >180 mmHg during screening). - Grand mal seizure within the last 6 months prior to screening. - Acute myocardial ischemia; hospitalization for congestive heart failure or myocardial infarction within 12 weeks before enrollment. - Stroke (hemorrhagic or ischemic) or transient ischemic attack within 12 weeks before enrollment. - Major surgery within 3 months prior to screening (excluding vascular access surgery). - Clinical evidence of systemic infection or inflammatory disease at the time of screening and up until enrollment.

For peritoneal dialysis subjects, an episode of peritonitis within 30 days before screening. - Known positivity for HIV antibody or Hepatitis B surface antigen.

Clinical evidence of current malignancy with the exception of basal cell or squamous cell carcinoma of the skin. - Blood transfusions within 8 weeks prior to screening or active bleeding. - Androgen therapy within 8 weeks prior to screening.

Systemic hematological disease (eg ,sickle cell anemia, myelodysplastic syndromes, hematological malignancy); myeloma; hemolytic anemia. - Other investigational products are excluded. - Subject is currently enrolled in, or has not yet completed, a period of at least 30 days since ending other investigational device or drug trial(s).

Psychiatric, addictive, or any other disorder that compromises ability to give truly informed consent for participation in this study. - Pregnant or breast feeding (women of child-bearing potential must be taking adequate contraceptive precautions). - Anticipating or scheduled for a living-related kidney transplant. - Known history of severe hyperparathyroidism (PTH >1500pg/ml) within 3 months prior top enrollment. - Currently receiving home hemodialysis treatment. - Currently receiving immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2005-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com